CLINICAL TRIAL: NCT06267638
Title: Comparison of Postoperative Pain Score Between Perioperative Intravenous Ketamine and Placebo in Patients Undergoing Unilateral Total Knee Arthroplasty Under General Anesthesia, A Prospective Randomized Controlled Trial Study
Brief Title: Comparison of Postoperative Pain Score Between Perioperative Intravenous Ketamine and Placebo in Patients Undergoing Unilateral Total Knee Arthroplasty Under General Anesthesia
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Ministry of Health, Thailand (Other Government)
Responsible Party: Principal Investigator, Numphung Sukantarat, Anesthsiologist of Chomthong hospital, Chiangmai, Ministry of Health, Thailand
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Chomthong hospital, Thailand
Record Dates: First submitted 2024-02-02; First posted 2024-02-20 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Knee Osteoarthritis
Keywords: ketamine; total knee arthroplasty; general anesthesia; Total Knee Arthropathy
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ketamine group (Experimental): Participant will receive intraoperative ketamine during total knee arthroplasty by Ketamine 0.5mg /kg loading then 0.25 mg/kg/hours until end of surgery
  Interventions: Drug: Ketamine group
- Placebo group (Placebo Comparator): Participant will receive intraoperative normal saline during total knee arthroplasty
  Interventions: Drug: Placebo group

INTERVENTIONS:
Drug: Ketamine group — Participants will receive intraoperative ketamine during total knee arthroplasty
  Arms: ketamine group
Drug: Placebo group — Participants will receive intraoperative normal saline during total knee arthroplasty
  Arms: Placebo group

SUMMARY:
The goal of this clinical trial is to compare postoperative pain score between perioperative intravenous ketamine and placebo in patients undergoing unilateral total knee arthroplasty under general anesthesia. The main question[s] it aims to answer are:

* Can perioperative intravenous ketamine reduce postoperative pain score during rest and movement at 0, 2, 4, 8, 12, 18, 24 hours better than no administration of Ketamine in patients undergoing Unilateral total knee arthroplasty under general anesthesia?
* Can perioperative intravenous ketamine reduce morphine consumption in postoperative 24 hours, length of hospital stay, first time to receive opioid and side effect or complication from ketamine and opioid better than no administration of Ketamine in patients undergoing Unilateral total knee arthroplasty under general anesthesia? Participants will receive intravenous ketamine intraoperative TKA and comparison group will receive placebo that is normal saline. Researchers will compare perioperative intravenous ketamine and placebo to see postoperative pain score, morphine consumption in postoperative 24 hours, length of hospital stay, first time to receive opioid and side effect or complication from ketamine and opioid.

ELIGIBILITY:
Inclusion Criteria:

1. A patient undergo unilateral total knee arthroplasty under General anesthesia at Chomthong Hospital Chiang Mai During 2024 to December 2025
2. Age is more than 18 years old
3. ASA (American society of anesthesiologist) status are I,I,III
4. A patient can cooperate in research

Exclusion Criteria:

* Patients allergic to local anesthetic agent
* Patient who has contraindication to use ketamine
* Patients has coagulopathy.
* Injection site is infected.
* Patients with chronic pain received painkillers for more than 3 months.
* The patient has a history of opioid use.
* The patient has a history of alcohol dependence.
* Patients allergic to fentanyl or morphine.
* Patient who has unstable cardiovascular disease
* Patient who has increase intracranial pressure and high ocular pressure
* Pregnancy
* The patient who has communication problems cannot describe the level of pain
* The patient refused to participate in the study.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-01-22 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain score at rest and movement | post operative time at 0 ,2 ,4 ,8 ,12 ,18 ,24 hours
  pain score at rest and movement by numeric rating scale 0-10

SECONDARY OUTCOMES:
First time to receive intravenous analgesic drug | First time to receive intravenous analgesic drug ( From finished anesthetic time until First time to receive intravenous analgesic drug(minute)
  First time to receive intravenous analgesic drug after operation was finished
Morphine consumption | post operative time at 0 ,2 ,4 ,8 ,12 ,18 ,24 hours
  Post operative morphine consumption or morphine equivalent (milligram)
Length of hospital stay | Time that patient was admited to hospital until patient was discharge from hospital.
  Length of hospital stay : When participant admit to discharge
side effect and complication from ketamine and opioid | post operative time within 24 hours
  Number of Participants with side effect form Ketamine and opioid: Hallucination, Nightmare, Arrythmia , Nausea vomiting respiratory distress ,Pruritus within 24 hours after operation. Do you have hallucination or nightmare? : yes no
  Nausea vomiting : - Severity of nausea 4 scale :
  0 = No
  1. =minimal nausea and vomiting don't need medication
  2. = nausea and vomiting participant was improved when received medication 3= nausea and vomiting participant wasn't improved when received medication Pruritus score 0= no
  1= minimal 2= severe and need medication respiratory distress : sedation scale 0 = awake
  1. minimal sedation : response to verbal conversation
  2. moderated sedation : sleeping but easy to response to verbal conversation
  3. deep sedation : difficult to response to

CONTACTS AND LOCATIONS:
Locations (1):
- Chomthong hospital, Chiang Mai, Thailand